CLINICAL TRIAL: NCT02656472
Title: A Pilot Study Comparing Anti-Inflammatory Effects Of Tranexamic Acid Versus Epsilon Aminocaproic Acid In Pediatric Congenital Heart Surgery
Brief Title: A Pilot Study Comparing Anti-Inflammatory Effects Of TXA Versus EACA In Pediatric Congenital Heart Surgery
Acronym: TXAEACA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: K5900283
Record Dates: First submitted 2015-12-29; First posted 2016-01-15 (Estimated); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Cardiac Surgery; Complication of Extracorporeal Circulation
Keywords: Pediatric Cardiac surgery; Inflammatory response; Tranexamic acid; Epsilon Aminocaproic Acid
MeSH Terms: interventions — Tranexamic Acid; Aminocaproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid Arm (Active Comparator): TXA arm will include 10 subjects who will receive TXA for duration of surgery.
  Interventions: Drug: Tranexamic acid
- Epsilon Aminocaproic Acid Arm (Active Comparator): EACA arm will include 10 subjects who will receive EACA for the duration of surgery.
  Interventions: Drug: Epsilon Aminocaproic Acid

INTERVENTIONS:
Drug: Tranexamic acid — TXA Loading dose: 31 mg/kg diluted to 2 ml/kg Normal saline (NS) -in syringe
  Other Names: TXA
  Arms: Tranexamic Acid Arm
Drug: Epsilon Aminocaproic Acid — Aminocaproic acid Loading dose: 75 mg/kg diluted to 2 ml/kg NS
  Other Names: EACA
  Arms: Epsilon Aminocaproic Acid Arm

SUMMARY:
The purpose of this study is to compare anti-inflammatory effects of two anti-fibrinolytic drugs (Tranexamic acid versus Epsilon-aminocaproic acid) in pediatric patients undergoing pediatric cardiac surgery.

DETAILED DESCRIPTION:
Bleeding under cardiopulmonary bypass (CPB) is one of the most common complications in patients undergoing pediatric cardiac surgery. The inflammatory response produced during and after CPB is a factor that adds significantly to the morbidity after cardiac surgery. A number of factors have been shown to be involved inducing the inflammatory response. These include complement system activation and activation of inflammatory cytokines, especially Interleukin (IL)-1, IL-6, IL-8 and Tumor necrosis factor (TNF) alpha.

Tranexamic Acid (TXA) and Epsilon-Aminocaproic Acid (EACA) are lysine analogues frequently used as anti-fibrinolytic agents in patients undergoing CPB. Many authors have highlighted the role of TXA in reducing blood loss and blood transfusion during and after CPB. Role of EACA and aprotinin in decreasing pro-inflammatory response during and after CPB has been well documented in adult literature. Patients undergoing redo sternotomy have higher inflammatory response as compared to patients undergoing first cardiac surgery. It has also been shown that the TXA can reduce the inflammatory response after CPB by acting directly or indirectly on the inflammatory cytokines.

There are no studies directly comparing the anti-inflammatory properties of EACA and TXA in the pediatric population undergoing CPB. In our institution, EACA is used as the standard of practice to reduce the blood loss during pediatric cardiac surgeries, but the investigators have now started using TXA more recently.

The aim of this study is to compare the anti-inflammatory and anti-fibrinolytic properties of these two anti-fibrinolytic agents in pediatric patients undergoing CPB for cardiac surgery.

Hypothesis: Tranexamic acid (TXA) has better anti-inflammatory profile as compared to €-Amino Caproic Acid (EACA) which may help in reducing blood loss, renal injury, hepatic injury and blood transfusion during and after CPB

Specific Objectives: During redo sternotomy procedures there is significant anti-inflammatory response which occurs and plays a role in increasing amount chest tube output, blood loss, renal injury, hepatic injury and ultimately patient morbidity and/or mortality. The proposed study will help to know if antifibrinolytic agents are beneficial in reducing the anti-inflammatory response produced and which of the two drugs (EACA or TXA), has a better anti-inflammatory profile when used in a similar setting for patients undergoing pediatric cardiothoracic surgery.

Specific Aims:

Evaluate whether TXA or EACA can decrease inflammatory response produced during redo sternotomy procedures in pediatric patients and which drug decreases the injury and/or cardiac dysfunction more as reflected by fluid balances, inotropic support, diuretic requirement, length of ventilator support, length of ICU stay, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pediatric cardiac surgery, with redo sternotomy needing cardiopulmonary bypass

Exclusion Criteria:

* Patients undergoing Fontan or Glenn procedures
* Allergy to EACA or TXA
* Baseline coagulation profile abnormality * (The coagulation profile will be used as an exclusion criteria, if results available. Occasionally the results of coagulation profile may be unavailable prior to surgery due to a clotted sample. For such patients, as per the current clinical practice, we would not be redrawing the lab solely for a research purpose)

  * Prothrombin time (PT) >50% of High Normal value
  * Partial Thromboplastin Time (PTT) > 50% of High Normal value
  * Platelets < 50,000/mm3
  * International normalized ratio (INR) >2
* Acute or chronic renal failure (creatinine > 2x high normal for age)
* Chronic hepatopathy (any transaminase > 2x high normal for age)
* Use of immunosuppressant drugs (within last 1 month)
* History of seizures (currently on antiepileptic drugs for epilepsy or history of seizure within last 6 months)

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew VanBergen, M.D., Principal Investigator — Director, Section of Pediatric Cardiac Critical Care
Locations (1):
- Advocate Childrens Hospital, Oak Lawn, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: From February 2016 to September 2016
Pre-assignment Details: 1 patient excluded after consent, prior to randomization, as exclusion criteria were present prior to surgery.
  At mid-study analysis, 1 significant outlier was noted (met inclusion criteria but was inpatient at time of randomization with multiple comorbidities where all other subjects were admitted on day of surgery).
Groups:
- Tranexamic Acid (TXA) Arm: TXA arm will include 10 subjects who will receive TXA for duration of surgery.
  Tranexamic acid: TXA Loading dose: 31 mg/kg diluted to 2 ml/kg NS
- Epsilon Aminocaproic Acid (EACA) Arm: EACA arm will include 10 subjects who will receive EACA for the duration of surgery.
  Epsilon Aminocaproic Acid: Aminocaproic acid Loading dose: 75 mg/kg diluted to 2 ml/kg NS.
Period: Overall Study
Arm/Group | Tranexamic Acid (TXA) Arm | Epsilon Aminocaproic Acid (EACA) Arm
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tranexamic Acid Arm: TXA arm included 10 subjects who received TXA for duration of surgery.
  TXA dosing strategy used an initial 31 mg/kg load at start of surgery, followed by 14 mg/kg/hr continuous infusion, and weight-dependent bolus dose after heparinization.
- Epsilon Aminocaproic Acid Arm: EACA arm included 10 subjects who will received EACA for the duration of surgery.
  EACA dosing strategy used an initial 75 mg/kg load at start of surgery, followed by 75 mg/kg/hr continuous infusion, and 75 mg/kg bolus dose after heparinization.
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Arm | Epsilon Aminocaproic Acid Arm | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (4.7) | 11.4 (6.0) | 10.5 (7.0)
Sex/Gender, Customized [Number; unit: participants]
  Male | 6 | 6 | 12
  Female | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: Weight (kg)] | 35.4 (19.2) | 11.4 (6.0) | 20.5 (22.2)
Height [Mean (Standard Deviation); unit: centimeters] | 136 (33.8) | 139 (38.0) | 137.5 (36.0)
STAT category [Mean (Standard Deviation); unit: units on a scale] — STAT Mortality Categories are a multi-institutional, validated complexity stratification tool for pediatric and congenital heart surgery. Operations were sorted by increasing risk and grouped into 5 categories (the STAT Mortality Categories). STAT Category 1 is associated with the lowest risk of mortality and STAT Category 5 is associated with the highest risk of mortality. The STAT Mortality Categories allow outcomes to be assessed in relation to the complexity of the operations being performed.
  units on a scale | 2.6 (1.0) | 2.4 (0.7) | 2.5 (0.85)

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Markers/Cytokines
Description: Consented patients had research-related blood draws (0.3 ml) at three time points: pre-CPB, post-CBP following protamine administration and 24 hours post-CPB. Average of the values run in duplicate was used for calculations. For samples with values reported as out of range (due to level being below detection), the lowest detectable value was assigned for analysis.
Time Frame: 24 hours post-surgery
Measure: Median (Inter-Quartile Range); unit: pg/dl
Groups:
- Tranexamic Acid (TXA) Arm: TXA dosing strategy used an initial 31 mg/kg load at start of surgery, followed by 14 mg/kg/hr continuous infusion, and weight-dependent bolus dose after heparinization.
- Epsilon Aminocaproic Acid (EACA) Arm: EACA dosing strategy used an initial 75 mg/kg load at start of surgery, followed by 75 mg/kg/hr continuous infusion, and 75 mg/kg bolus dose after heparinization.
Arm/Group | Tranexamic Acid (TXA) Arm | Epsilon Aminocaproic Acid (EACA) Arm
Number analyzed (Participants) | 10 | 10
pg/dl
  Pre-CPB IL-1B | 1.5 [0.8 to 1.8] | 2.1 [1.4 to 3.5]
  Pre-CPB-IL2 | 1.6 [1.1 to 2.2] | 2.2 [1.4 to 4.3]
  Pre-CPB-IL4 | 0.4 [0.2 to 0.6] | 0.6 [0.2 to 1.1]
  Pre-CPB-IL5 | 0.2 [0.1 to 0.4] | 0.4 [0.2 to 0.9]
  Pre-CPB-IL6 | 0.2 [0.1 to 1.5] | 0.6 [0.2 to 1.1]
  Pre-CPB-IL8 | 3.0 [1.8 to 6.6] | 6.1 [2.2 to 13.1]
  Pre-CPB IL-10Beta | 3.0 [2.3 to 6.0] | 3.2 [2.2 to 6.5]
  Pre-CPB IL-12 | 0.2 [0.2 to 0.5] | 0.4 [0.2 to 2.6]
  Pre-CPB IL-13 | 0.2 [0.0 to 1.5] | 1.3 [0.0 to 7.8]
  Pre-CPB TNF Alpha | 16.6 [12.7 to 24.0] | 19.6 [10.9 to 32.5]
  Pre-CPB IFN gamma | 1.1 [1.1 to 1.8] | 1.0 [0.3 to 3.2]
  Pre-CPB GM-CSF | 3.6 [2.7 to 6.7] | 5.4 [2.1 to 11.0]
  Pre-CPB MCP-1 | 184.7 [133 to 228.6] | 224.6 [170.7 to 323.4]
  Post-CPB IL-1 | 1.5 [1.2 to 1.6] | 2.2 [1.2 to 5.4]
  Post-CPB IL-2 | 2.2 [1.7 to 2.5] | 2.7 [1.5 to 4.1]
  Post-CPB IL-4 | 0.4 [0.2 to 0.6] | 0.6 [0.2 to 3.7]
  Post-CPB IL-5 | 0.1 [0.1 to 0.3] | 0.3 [0.1 to 1.6]
  Post-CPB IL-6 | 43.0 [19.6 to 69.6] | 28.5 [21.9 to 30.9]
  Post-CPB IL-8 | 19.6 [12.3 to 69.7] | 28.0 [11.3 to 57.8]
  Post-CPB IL-10 | 1047.6 [646.4 to 1996.8] | 2338.3 [1995.5 to 2839.3]
  Post-CPB IL-12 | 0.2 [0.2 to 1.9] | 0.9 [0.2 to 3.9]
  Post-CPB IL-13 | 0.2 [0.0 to 0.7] | 1.4 [0.0 to 15.1]
  Post-CPB TNF Alpha | 15.3 [11.5 to 22.8] | 15.2 [9.6 to 27.6]
  Post-CPB IFN Gamma | 1.1 [0.1 to 2.1] | 0.9 [0.1 to 2.7]
  Post-CPB GM-CSF | 5.8 [3.9 to 8.4] | 7.3 [5.3 to 13.0]
  Post-CPB MCP-1 | 308.6 [256.4 to 507.9] | 251.9 [218.6 to 385.5]
  24 hour post CPB IL-1 | 1.2 [0.9 to 1.8] | 1.0 [1.0 to 2.6]
  24 hour post CPB IL-2 | 1.3 [0.9 to 2.2] | 1.4 [0.8 to 3.4]
  24 hour post CPB IL-4 | 0.6 [0.2 to 0.6] | 0.6 [0.2 to 0.8]
  24 hour post CPB IL-5 | 0.1 [0.0 to 0.5] | 0.0 [0.0 to 0.6]
  24 hour post CPB IL-6 | 14.7 [8.3 to 44.0] | 28.0 [10.8 to 39.6]
  24 hour post CPB IL-8 | 7.5 [5.1 to 39.7] | 10.9 [9.1 to 21.8]
  24 hour post CPB IL-10 | 6.2 [4.5 to 33.3] | 13.3 [5.5 to 27.2]
  24 hour post CPB IL-12 | 0.2 [0.2 to 0.4] | 0.2 [0.2 to 2.8]
  24 hour post CPB IL-13 | 0.1 [0.0 to 0.9] | 0.6 [0.0 to 5.7]
  24 hour post CPB TNF Alpha | 10.8 [8.3 to 16.1] | 13.2 [8.1 to 16.3]
  24 hour post CPB IFN Gamma | 0.6 [0.3 to 0.6] | 1.0 [0.3 to 2.3]
  24 hour post CPB GM-CSF | 5.1 [3.1 to 8.8] | 5.1 [1.6 to 9.5]
  24 hour post MCP-1 | 180.0 [92.3 to 235.0] | 180.2 [09.8 to 221.1]

2. Secondary Outcome: Chest Tube Output
Description: Chest tube output in ml/kg for the first 48 hours
Time Frame: 48 hours post-surgery
Measure: Median (Inter-Quartile Range); unit: ml/kg
Groups:
- Tranexamic Acid Arm: TXA dosing strategy used an initial 31 mg/kg load at start of surgery, followed by 14 mg/kg/hr continuous infusion, and weight-dependent bolus dose after heparinization.
- Epsilon Aminocaproic Acid Arm: EACA dosing strategy used an initial 75 mg/kg load at start of surgery, followed by 75 mg/kg/hr continuous infusion, and 75 mg/kg bolus dose after heparinization.
Arm/Group | Tranexamic Acid Arm | Epsilon Aminocaproic Acid Arm
Number analyzed (Participants) | 10 | 10
ml/kg | 5.1 [3.7 to 18.4] | 7.8 [6.1 to 16.7]

3. Secondary Outcome: Blood Replacement Volume
Description: Compare the volume of blood product replacement needed in first 48 hours of surgery (including blood products used in OR)
Time Frame: 48 hours post-surgery
Measure: Median (Inter-Quartile Range); unit: ml/kg
Groups:
- TXA Group: TXA dosing strategy used an initial 31 mg/kg load at start of surgery, followed by 14 mg/kg/hr continuous infusion, and weight-dependent bolus dose after heparinization.
- EACA Group: EACA dosing strategy used an initial 75 mg/kg load at start of surgery, followed by 75 mg/kg/hr continuous infusion, and 75 mg/kg bolus dose after heparinization.
Arm/Group | TXA Group | EACA Group
Number analyzed (Participants) | 10 | 10
ml/kg
  pRBC | 0.0 [0.0 to 8.7] | 0.0 [0.0 to 12.7]
  Platelets | 2.0 [0.0 to 7.5] | 1.4 [0.0 to 8.3]
  FFP | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 5.6]

4. Secondary Outcome: Platelet Levels
Description: Antifibrinolytic effect using platelets levels x 1000/mL
Time Frame: Immediately post-surgery and 24 hours post-surgery
Measure: Mean (Standard Deviation); unit: Platelets x1000/mL
Arm/Group | TXA Group | EACA Group
Number analyzed (Participants) | 10 | 10
Platelets x1000/mL
  Platelet Day 0 | 163.7 (58.2) | 185.1 (54.5)
  Platelet Day 1 | 124.8 (47.8) | 162.8 (49.4)

5. Secondary Outcome: Liver Enzymes
Description: Tests were recorded and compared between the groups to analyze the effect of the antifibrinolytic agent used on the amount of blood loss as well as effect of inflammation on the liver and kidney.
Time Frame: Immediately post-surgery and 24 hours post-surgery
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tranexamic Acid Arm | Epsilon Aminocaproic Acid Arm
Number analyzed (Participants) | 10 | 10
U/L
  AST Day 0 | 131.8 (130.8) | 119.3 (162.4)
  AST Day 1 | 254.8 (307.8) | 175.1 (225.7)
  ALT Day 0 | 36.6 (24.2) | 74.5 (122.3)
  ALT Day 1 | 29.7 (13.9) | 31.4 (14.5)

6. Secondary Outcome: Hemoglobin
Description: as for outcome 5
Time Frame: Immediately post-surgery and 24 hours post-surgery
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Tranexamic Acid Arm | Epsilon Aminocaproic Acid Arm
Number analyzed (Participants) | 10 | 10
g/dl
  Hemoglobin Day 0 | 10.2 (1.7) | 11.1 (1.8)
  Hemoglobin Day 1 | 10.3 (1.3) | 9.9 (1.7)

7. Secondary Outcome: Creatinine
Description: as for outcome 5
Time Frame: Immediately post-surgery and 24 hours post-surgery
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Tranexamic Acid Arm | Epsilon Aminocaproic Acid Arm
Number analyzed (Participants) | 10 | 10
mg/dl
  creatinine Day 0 | 0.6 (0.2) | 0.6 (0.2)
  creatinine Day 1 | 0.5 (0.1) | 0.7 (0.2)

8. Secondary Outcome: Length of Stay
Description: Length of stay in the ICU and overall hospital stay.
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tranexamic Acid Arm | Epsilon Aminocaproic Acid Arm
Number analyzed (Participants) | 10 | 10
days
  ICU length of stay | 4.0 [2.0 to 5.5] | 2.0 [1.8 to 4.0]
  Hospital length of stay | 4.0 [2.0 to 5.8] | 3.5 [2.0 to 12.5]

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Tranexamic Acid Arm: TXA arm will include 10 subjects who will receive TXA for duration of surgery.
  Tranexamic acid: TXA Loading dose: 31 mg/kg diluted to 2 ml/kg NS.
Arm/Group | Tranexamic Acid Arm | Epsilon Aminocaproic Acid Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid Arm (N=10) | Epsilon Aminocaproic Acid Arm (N=10)
Pulmonary hemorrage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — 1 patient had acute pulmonary hemorrhage noted 36 hours after surgery, requiring reintubation. The likely etiology was spontaneous rupture of tracheobronchial vessel and was felt to be unrelated to TXA use.

LIMITATIONS AND CAVEATS:
Small sample size and wide age range lead to substantial variation in values, making it difficult to draw conclusions. Biomarker levels were collected at three time points, not including a 4-hour post-CPB level, when most cytokines are known to peak.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02656472/Prot_SAP_000.pdf